CLINICAL TRIAL: NCT03488459
Title: Influence of Preoperative Support on Anxiety, Pain and Satisfaction With Postoperative Analgesia in Children and Adolescents After Thoracic Surgeries: a Randomized Double Blind Study
Brief Title: Influence of Preoperative Support on Anxiety, Pain and Satisfaction With Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute for Tuberculosis and Lung Diseases, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10.5
Record Dates: First submitted 2018-03-22; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Pain, Postoperative; Surgery, Thoracic
Keywords: anxiety; preoperative education; psychologist; thoracotomy; Ravitch procedure; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine preoperative information from a nurse (Other)
  Interventions: Behavioral: Routine preoperative information from a nurse
- Additional information support from a psychologist (Experimental)
  Interventions: Behavioral: Additional information support from a psychologist

INTERVENTIONS:
Behavioral: Routine preoperative information from a nurse — Routine preoperative information from a nurse.
  Arms: Routine preoperative information from a nurse
Behavioral: Additional information support from a psychologist — Routine preoperative information from a nurse + additional information support from a psychologist.
  Arms: Additional information support from a psychologist

SUMMARY:
The aim of this study was to analyze a relationship between information support provided by an interdisciplinary team and the levels of anxiety, pain and satisfaction with postoperative analgesia in children and adolescents subjected to thoracic surgeries.

DETAILED DESCRIPTION:
The study included 112 consecutive pediatric patients qualified for lateral thoracotomy or Ravitch procedure. The subjects were randomized to the control group (n=56) provided with a routine preoperative information from a nurse, and the experimental group (n=56) offered additional psychological consultation.

ELIGIBILITY:
Inclusion Criteria:

* thoracic surgery (lateral thoracotomy or Ravitch procedure),
* the American Society of Anesthesiologists score 1 or 2.

Exclusion Criteria:

* presence of a mental disorder,
* anticancer treatment,
* preoperative pain,
* problems with verbal communication ,
* lack of postoperative drainage of the chest.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
Change in anxiety intensity scores | day prior to surgery, postoperative day 2
  Anxiety was determined with a Polish version of the self-inventory, either for children between 9 and 14 years of age, i.e. State-Trait Anxiety Inventory for Children (STAI-C; range: 20-60 pts) or for adolescents, i.e. State-Trait Anxiety Inventory (STAI; range: 20-80 pts). The instrument consisting of two separate 20-item scales measuring state and trait anxiety. In this study, the levels of anxiety were determined twice: one day prior to surgery (both trait and state anxiety) and 48 h after the procedure (only state anxiety). The results were expressed as sten scores, from 1-10 (1-4 = low level of anxiety, 5-6 = moderate level of anxiety, >7 = high level of anxiety).

SECONDARY OUTCOMES:
Pain intensity scores at rest | postoperative hours: 1, 2, 4, 11, 24, 48
  The Numeric Rating Scale (NRS) was used to evaluate the intensity of pain, where 0 meant no pain, and 10 - the most severe pain.
Pain intensity scores during deep breathing | postoperative hours: 1, 2, 4, 11, 24, 48
  The Numeric Rating Scale (NRS) was used to evaluate the intensity of pain, where 0 meant no pain, and 10 - the most severe pain.
Pain intensity scores during coughing | postoperative hours: 1, 2, 4, 11, 24, 48
  The Numeric Rating Scale (NRS) was used to evaluate the intensity of pain, where 0 meant no pain, and 10 - the most severe pain.
Patient satisfaction | postoperative day 2
  Satisfaction was evaluated on a 4-item scale: analgesia was rated as insufficient, poor, good or very good

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Tuberculosis and Lung Diseases, Pediatric Division, Rabka-Zdrój, Małopolska, Poland

REFERENCES:
- [Background] Chieng YJ, Chan WC, Klainin-Yobas P, He HG. Perioperative anxiety and postoperative pain in children and adolescents undergoing elective surgical procedures: a quantitative systematic review. J Adv Nurs. 2014 Feb;70(2):243-55. doi: 10.1111/jan.12205. Epub 2013 Jul 19. PMID 23865442
- [Background] Cuzzocrea F, Gugliandolo MC, Larcan R, Romeo C, Turiaco N, Dominici T. A psychological preoperative program: effects on anxiety and cooperative behaviors. Paediatr Anaesth. 2013 Feb;23(2):139-43. doi: 10.1111/pan.12100. PMID 23289773
- [Background] Fincher W, Shaw J, Ramelet AS. The effectiveness of a standardised preoperative preparation in reducing child and parent anxiety: a single-blind randomised controlled trial. J Clin Nurs. 2012 Apr;21(7-8):946-55. doi: 10.1111/j.1365-2702.2011.03973.x. Epub 2012 Feb 3. PMID 22300416
- [Derived] Tomaszek L, Cepuch G, Fenikowski D. Influence of preoperative information support on anxiety, pain and satisfaction with postoperative analgesia in children and adolescents after thoracic surgery: A randomized double blind study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2019 Jun;163(2):172-178. doi: 10.5507/bp.2018.060. Epub 2018 Oct 5. PMID 30305761